CLINICAL TRIAL: NCT04582903
Title: Send-In Sample Collection for Comprehensive Analyses of Innate and Adaptive Immune Responses During Acute Infections With, and Convalescence From, Emerging or Re-emerging Respiratory Viruses
Brief Title: Send-In Sample Collection for Comprehensive Analyses of Innate and Adaptive Immune Responses During Acute COVID-19 and Convalescence
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000044; 000044-I
Record Dates: First submitted 2020-10-09; First posted 2020-10-12 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-13

CONDITIONS: COVID-19 Infection
Keywords: severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); Repository; Pandemic; Genetics; Proteomics; Natural History
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Biological Relative: Biological relative of a participant being studied under this protocol. Relatives may be biological mother, father, siblings, children, grandparents, aunts, uncles, or first cousins
- Confirmed or Suspected SARS-CoV-2 infection: Patient with a known or suspected diagnosis of SARS-CoV-2 infection (past or current), typically but not always supported by a positive PCR test for viral RNA
- Exposed but Uninfected: Individual who has remained uninfected with negative SARS-CoV-2 serologies despite heavy or extensive COVID-19 exposure in the workplace or home environment

SUMMARY:
Background:

Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) causes coronavirus disease 2019 (COVID-19). The global outbreak of COVID-19 is a major public health problem. COVID-19 causes a wide range of symptoms. These symptoms range from mild breathing problems to life-threatening problems or death. Some people have no symptoms. This study aims to learn how acute and late immune responses to COVID-19 lead to different outcomes. The immune system is the body s defense against germs, including viruses, that invade the body.

Objective:

To characterize the immune responses during and after SARS-CoV-2 infection and determine if there is any relationship to clinical course and outcome.

Eligibility:

People ages 0 99 who have confirmed or suspected SARS-CoV-2 infection, people who are not infected despite heavy exposure, and relatives of enrolled participants.

Design:

This is a sample collection protocol to receive send-in biological specimens for exploratory studies, including gene testing. Participants will not be seen at the NIH for study visits.

Study staff will talk with participants health care providers to screen them for the study. Participants enrolled into the protocol will send samples and clinical information at least once and more often if the participant has COVID-19. All participants will provide blood samples and possibly stool. We may also ask for left over specimens from any medical procedures completed as part of medical care. The study staff will also request participants health care providers to complete a survey to collect demographic and medical data. Some of this information may need to be provided directly by the participant.

Pregnant individuals are invited to participate and may be asked to give cord blood samples after delivery. Study findings that affect participants health may be shared with their health care provider. Depending on findings, participants may be contacted to take part in other NIH studies.

DETAILED DESCRIPTION:
Study Description:

This is a prospective sample collection protocol to receive send-in biological samples (e.g., blood, saliva, stool, urine, and leftover clinically collected samples) for exploratory studies to characterize the immune response to coronavirus disease 2019 (COVID-19) or other emerging or re-emerging respiratory viruses. Participants will not be seen at the NIH for study visits. Under this protocol, samples will be collected longitudinally from patients with confirmed or suspected severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection or other emerging or re-emerging respiratory viruses and sent to the NIH for research evaluations. Additionally, samples will be collected from uninfected patients and patient relatives. Testing will be performed to improve understanding of host immune responses to these viruses, including but not limited to genetic, molecular, and proteomic testing. Findings relevant to participants' health and medical care may be returned to them and their referring health care providers or study teams.

Objectives:

Primary Objective:

To achieve genetic, immunologic, molecular, and virologic characterization of the host immune responses during and after infection with SARS-CoV-2 or other emerging or re-emerging respiratory viruses, which will be correlated with clinical course and outcome data.

Endpoints:

Primary Endpoints:

1. Identification of genetic variants that are associated with either severe/lethal disease or resistance to infection with SARS-CoV-2 or other emerging or re-emerging respiratory viruses.
2. Characterization of the dynamic changes of innate and adaptive immune responses acutely and during convalescence after infection with SARS-CoV-2 or other emerging or re-emerging respiratory viruses.
3. Measurement of proinflammatory/anti-inflammatory cytokines, including the interferon (IFN) signature response, produced acutely and during convalescence after infection with SARS-CoV-2 or other emerging or re-emerging respiratory viruses.
4. Characterization of serological responses against SARS-CoV-2, other viruses or microbiota, and host antigens.
5. Survey of other potential blood proteomic biomarkers of disease.
6. Characterization of intrapatient SARS-CoV-2 or other emerging or re-emerging virus genetic variation and evolution during infection and convalescence.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants enrolled onto this protocol must meet all of the following criteria:

1. Aged 0-99 years (including viable neonates).
2. Meets one of the following criteria:

   1. Patient with a known or suspected diagnosis of infection (past or current) with SARS-CoV-2 or an emerging or re-emerging respiratory virus, typically but not always supported by a positive PCR test for viral RNA;
   2. Individual who has remained uninfected with negative virus serologies despite heavy or extensive exposure to the emerging or re-emerging respiratory virus in the workplace or home environment; or
   3. Biological relative of a participant being studied under this protocol. Relatives may be biological mother, father, siblings, children, grandparents, aunts, uncles, or first cousins.
3. For individuals considered for enrollment as uninfected individuals and biological relatives, able to provide informed consent.
4. Willing to allow genetic testing.
5. Willing to allow storage of samples and data for future research.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

1. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Since patients can be concurrently infected with multiple respiratory viruses, positive testing for other viruses such as rhinovirus, influenza virus, etc., does not exclude an individual from study participation where there remains a high clinical suspicion of infection with the emerging or re-emerging respiratory virus of interest despite negative testing for it.

Co-enrollment guidelines: Participants may be co-enrolled in other studies; however, study staff should be notified of co-enrollment.

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We plan to enroll up to 500 total participants in this protocol, including up to 300 patients with SARS-CoV-2 infection and 200 other participants (patient relatives and individuals who remain uninfected despite heavy or extensive COVID-19 exposure in the workplace or home environment). Health care providers worldwide will contact the study staff to request enrollment of patients and/or their relatives. Additionally, investigators may refer patients from other clinical studies.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
Characterization of the dynamic changes of innate and adaptive immune responses during SARS CoV 2 infection and convalescence. | End of Study
  These endpoints were chosen to provide in depth molecularmeasurements of a wide variety of innate and adaptive host immuneresponses to a novel pathogen in heterogenous patients. This is anexploratory hypothesis generating study to identify findings for validation in future studies. These endpoints are needed to better understand pathogenic mechanisms, improve prognostic tools, optimize existing therapies, and identify new targets for treatment.
Identification of genetic variants that are associated with either severe/lethal COVID-19 or resistance to SARS CoV 2 infection. | End of Study
  These endpoints were chosen to provide in depth molecular measurements of a wide variety of innate and adaptive host immune responses to a novel pathogen in heterogenous patients. This is an exploratory hypothesis generating study to identify findings for validation in future studies. These endpoints are needed to better understand pathogenic mechanisms, improve prognostic tools, optimize existing therapies, and identify new targets for treatment.
Measurement of proinflammatory/anti inflammatory cytokines produced during SARS CoV 2 infection and convalescence, including the IFN signature response. | End of Study
  These endpoints were chosen to provide in depth molecular measurements of a wide variety of innate and adaptive host immune responses to a novel pathogen in heterogenous patients. This is an exploratory hypothesis generating study to identify findings for validation in future studies. These endpoints are needed to better understand pathogenic mechanisms, improve prognostic tools, optimize existing therapies, and identify new targets for treatment.
Survey of other potential blood proteomic biomarkers of disease. | End of Study
  These endpoints were chosen to provide in depth molecular measurements of a wide variety of innate and adaptive host immune responses to a novel pathogen in heterogenous patients. This is an exploratory hypothesis generating study to identify findings for validation in future studies. These endpoints are needed to better understand pathogenic mechanisms, improve prognostic tools, optimize existing therapies, and identify new targets for treatment.
Characterization of serological responses against SARS CoV 2, other viruses or microbiota, and host antigens. | End of Study
  These endpoints were chosen to provide in depth molecular measurements of a wide variety of innate and adaptive host immune responses to a novel pathogen in heterogenous patients. This is an exploratory hypothesis generating study to identify findings for validation in future studies. These endpoints are needed to better understand pathogenic mechanisms, improve prognostic tools, optimize existing therapies, and identify new targets for treatment.
Characterization of intrapatient SARS-CoV-2 genetic variation and evolution during infection and convalescence. | End of Study
  These endpoints were chosen to provide in depth molecular measurements of a wide variety of innate and adaptive host immune responses to a novel pathogen in heterogenous patients. This is an exploratory hypothesis generating study to identify findings for validation in future studies. These endpoints are needed to better understand pathogenic mechanisms, improve prognostic tools, optimize existing therapies, and identify new targets for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Su, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Niaid/Lcim, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
This study is part of a multi-institute project at the NIH and we may share de-identified information to the various participating institutes and investigators as needed.

REFERENCES:
- [Background] Casanova JL, Su HC; COVID Human Genetic Effort. A Global Effort to Define the Human Genetics of Protective Immunity to SARS-CoV-2 Infection. Cell. 2020 Jun 11;181(6):1194-1199. doi: 10.1016/j.cell.2020.05.016. Epub 2020 May 13. PMID 32405102
- [Background] Burbelo PD, Riedo FX, Morishima C, Rawlings S, Smith D, Das S, Strich JR, Chertow DS, Davey RT, Cohen JI. Sensitivity in Detection of Antibodies to Nucleocapsid and Spike Proteins of Severe Acute Respiratory Syndrome Coronavirus 2 in Patients With Coronavirus Disease 2019. J Infect Dis. 2020 Jun 29;222(2):206-213. doi: 10.1093/infdis/jiaa273. PMID 32427334
- [Background] Gabutti G, d'Anchera E, Sandri F, Savio M, Stefanati A. Coronavirus: Update Related to the Current Outbreak of COVID-19. Infect Dis Ther. 2020 Jun;9(2):241-253. doi: 10.1007/s40121-020-00295-5. Epub 2020 Apr 8. PMID 32292686